CLINICAL TRIAL: NCT06501144
Title: Real-world Longitudinal Follow-up Study of a Digital Health Application in Erectile Dysfunction
Acronym: RELOED
Status: Completed | Type: Observational
Sponsor: Kranus Health GmbH (Industry)
Collaborators: Centre of Reproductive Medicine and Andrology, department of Clinical and Surgical Andrology, Münster (Unknown)
Responsible Party: Sponsor
Other Study IDs: RELOED01
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Erectile Dysfunction; Sexual Dysfunction
Keywords: Erectile Dysfunction; Digital Health; App-based Therapy; Digital Therapeutics; Real World Evidence; Mobile Health; Behavioral Interventions; Quality of Life; Lifestyle Changes; Urology
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the long-term effectiveness of a digital health application for treating erectile dysfunction in men aged 18 and older. The main questions it aims to answer are:

* Will participants maintain an improvement of their erectile function, that means maintain an improvement of at least 3 points in the IIEF-5 score at 3 months post-therapy?
* How does the application affect overall health status and disease-related quality of life?

Participants will:

* Complete validated questionnaires (IIEF-5, PGI-I, QOL-Med) to track erectile function, overall health status, and quality of life at up to two follow-up points after using the app with a 3-month self-management program combining cardiovascular training, pelvic floor exercises, psychological support, and educational content.
* Provide information on demographics, risk factors, and other relevant health characteristics for subgroup analysis.

DETAILED DESCRIPTION:
The intervention that needs to be completed prior participation in this study involves a digital therapy program delivered via a smartphone or tablet application. This program includes several components aimed at addressing different aspects for the treatment of erectile dysfunction:

* Pelvic Floor Exercises
* Cardiovascular Exercises
* Physiotherapeutic Exercises
* Mental or sexual therapeutic Exercises
* Educational Content

Overall, the digital therapy program is designed to provide comprehensive support for men with erectile dysfuntion, addressing both physical and psychological aspects of the condition to improve symptom severity, quality of life, and patient activation.

ELIGIBILITY:
Inclusion Criteria:

* Men with erectile dysfunction of organic origin (ICD 10 code N48.4) and IIEF-5 score < 21 as determined at therapy start with Kranus EDERA
* Completion of the 12-week app-based therapy with Kranus EDERA
* Improvement in the IIEF-5 score of ≥ 3 points after completion of the Kranus EDERA therapy compared to the score at the start of the therapy
* Age over 18

Exclusion Criteria:

* Failure to provide informed consent
* Started a new therapy with Kranus EDERA between the end of the last therapy cycle and patient survey
* Started PDE-5 inhibitor treatment during the Kranus EDERA therapy or between the end of the last therapy cycle and patient survey
* Underwent prostatectomy (removal of the prostate gland), radiation or seeds of the prostate gland during the Kranus EDERA therapy or between the end of the last therapy cycle and patient survey
* Performed auto-injection therapy (SKAT, MUSE) during the Kranus EDERA therapy or between the end of the last therapy cycle and patient survey
* Obtained a penile implant during the Kranus EDERA therapy or between the end of the last therapy cycle and patient survey
* Underwent major surgery in the small pelvis with probable impairment of the neurovascular supply (e.g., rectum resection, urinary bladder removal) during the Kranus EDERA therapy or between the end of the last therapy cycle and patient survey
* Nervous diseases (e.g., multiple sclerosis (MS), Parkinson's disease, stroke, dementia, psychiatric diseases) acquired during the Kranus EDERA therapy or between the end of the last therapy cycle and patient survey
* Developed pronounced circulatory disorders (peripheral arterial occlusive disease) during the Kranus EDERA therapy or between the end of the last therapy cycle and patient survey
* Trauma involving the pelvis/penis/spine during the Kranus EDERA therapy or between the end of the last therapy cycle and patient survey
* Any other newly developed diseases potentially affecting erectile function (e.g., leading to a longer period of hospitalization) during the Kranus EDERA therapy or between the end of the therapy cycle and patient survey

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Because this study investigates the effects of a therapy program on erectile dysfunction, eligibility requires participants to have male primary genital anatomy, regardless of gender identity.
Study Population: This study will include adults with erectile dysfunction who have started the 3-month therapy with the app-based therapeutic within the last 6 months
Sampling Method: Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Assessment of the real-world longitudinal effect of the intervention | 6 months after start of the app-based therapy
  The primary endpoint is the rate of patients maintaining an IIEF-5 score improvement of ≥ 3 points compared to baseline (start of app-based therapy) after the app-based therapy

SECONDARY OUTCOMES:
Assessment of the real-world effect of the intervention on overall improvement of patients' health status | 6 months after start of the app-based therapy
  Assessment of overall improvement of patients' health status using the PGI-I questionnaire
Assessment of the real-world effect of the intervention on disease-related quality of life | 6 months after start of the app-based therapy
  Assessment of disease-related quality of life using the QOL-Med questionnaire

OTHER OUTCOMES:
Other outcome measures/variables | 6 months after start of the app-based therapy
  * Demographics and patient characteristics (specified in the study protocol)
  * IIEF-5
    •. PGI-I
  * QOL-MED
  * BMI changes
  * Responders (A priori responder definition of patients with the minimal important difference (MID) of an ≥ 3 points IIEF-5 score improvement to assess the maintenance of a therapeutic effect according to the hypothesis this study aims to investigate)
  Derived variables
  * Changes of IIEF-5 from baseline
  * Changes of IIEF-5 from baseline
  * Changes of IIEF-5 from end of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Kliesch, MD, Principal Investigator — CeRA Münster, Centre of Reproductive Medicine and Andrology , department of Clinical and Surgical Andrology, Münster, Germany
Locations (1):
- CeRa Münster, Centre of Reproductive Medicine and Andrology, Münster, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wiemer L, Bartelheimer T, Raschke R, Miller K. [First data from a digital health app for erectile dysfunction]. Urologie. 2022 Sep;61(9):971-981. doi: 10.1007/s00120-022-01872-x. Epub 2022 Jun 20. German. PMID 35925101
- [Background] Kliesch S, Cremers JF, Krallmann C, Epplen R, Scheffer B, Schubert T, Schubert M, Dreger NM, Raschke R, Khaljani E, Maxeiner A, Miller K, Wiemer L, Zitzmann M. App-based Therapy of Erectile Dysfunction Using a Digital Health Application (EDDIG Study): A Randomized, Single-blind, Controlled Trial. Eur Urol Focus. 2024 Dec;10(6):1003-1010. doi: 10.1016/j.euf.2024.05.020. Epub 2024 Jun 8. PMID 38853028